CLINICAL TRIAL: NCT06650371
Title: Comparative Study Between the Performance of Opioid Free Anesthesia Versus Conventional Opioid Based Anesthesia Regarding Achievement of Enhanced Recovery in Laparoscopic Bariatric Surgeries
Brief Title: Opioid Free Anesthesia Versus Opioid Based Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eman Mohamed Zain Eldeen, Doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD126/2024
Record Dates: First submitted 2024-09-29; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Opioid Free Anesthesia; Laparoscopic Bariatric Surgeries
Keywords: Opioid free anesthesia; laparoscopic bariatric surgeries

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fentanyl infusion (Active Comparator): Analgesia will be offered by fentanyl in induction and maintenance according to ideal body weight (IBW).
  Interventions: Drug: Fentanyl infusion
- Dexamedomedine and ketamine infusion (Active Comparator): Opioid free anesthesia Analgesia will be offered by syringe containing ketamine and dexmedetomidine in induction and maintenance according to IBW.
  Interventions: Drug: Dexamedomedine and ketamine infusion

INTERVENTIONS:
Drug: Fentanyl infusion — opioid based anesthesia analgesia will be offered by fentanyl in induction and maintenance according to Ideal Body Weight (IBW).
  Arms: Fentanyl infusion
Drug: Dexamedomedine and ketamine infusion — Analgesia will be offered by syringe containing ketamine and Dexmedetomidine in induction and maintenance according to IBW.
  Arms: Dexamedomedine and ketamine infusion

SUMMARY:
This Study aims to evaluate the efficacy of opioid free general anesthesia in achieving enhanced recovery after surgery (ERAS) in laparoscopic bariatric surgery in terms of post-operative recovery time, cumulative pethidine consumption and number of episodes of postoperative nausea and vomiting(PONV).

DETAILED DESCRIPTION:
While opioids have been commonly used in the operating room due to their effectiveness in pain management and anesthesia, there are numerous common side effects that have an impact on patient recovery. Obese patients or those with pre-existing respiratory difficulties such as sleep apnea or chronic obstructive pulmonary disease are more likely to experience respiratory failure after getting opiate therapy. Other effects of opioid use include gastro-intestinal obstacles such nausea, vomiting, and constipation.

The concept of opioid-free anesthesia evolved due to the potential adverse side effects associated with intraoperative opioid usage.

This study examines nociceptive monitoring's potential role in opioid-free anesthesia, as well as research on the topic. This study aims to compare the effects of an opioid-free anesthesia (OFA) regimen versus an opioid-based anesthesia (OBA) regimen on postoperative pain and enhanced recovery in patients undergoing bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a scheduled laparoscopic bariatric surgery under general anesthesia.
* Age group: 18-65 years old.
* BMI greater than 35 to 50 Kg/m2
* ASA physical status classes I and II.

Exclusion Criteria:

* Patient refusal.
* ASA physical status classes III and IV.
* Anticipated difficult intubation.
* Hypersensitivity to any drugs used in this study. Inability to extubate the patient at the end of the operation. Conversion to laparotomy. Patients for whom the anesthetic regimen is changed intraoperatively (from OFA to OBA or vice versa).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Time between the end of analgesic used and an Aldrete score > 9 (when applicable). | 15 minutes
  Decrease opioid usage ,decrease recovery time
Time between the end of operation to PACU | 15 minutes
  Decrease opioid usage ,decrease recovery time

SECONDARY OUTCOMES:
Cumulative pethidine consumption | 24 hours postoperative
  decrease the need to postoperative pethidine
Number of episodes of nausea and vomiting [Time Frame: During the 24 hours following extubation]. | 24 hours postoperative
  number of episodes of nausea and vomiting postoperative